CLINICAL TRIAL: NCT01263041
Title: Effect of Early Enteral Supplementation of L-arginine and Glutamine on Preterm Neonate
Brief Title: Effect of L-arginine and Glutamine on Preterm
Acronym: preterm
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, ghada saleh, G. Saleh, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ghada a. saleh MD protocol
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: NEC; Sepsis
Keywords: Glutamine, NEC, L-arginine,Preterm,Sepsis
MeSH Terms: conditions — Sepsis; Enterocolitis, Necrotizing | interventions — Glutamine; Arginine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- glutamine, PT, sepsis (Experimental): enteral or via NG tube dose of 312mg/kg/day divided every 12 hours from starting feeding up to 30 says post natal age + usual care and medications
  Interventions: Drug: Glutamine
- Control (No Intervention): after been allocated, will receive nothing and observed for the same outcomes
- L-arginine,NEC, PT (Experimental): enteral or via NG tube dose of 260 mg/kg/day divided every 12 hours from starting feeding up to 30 says post natal age + usual care and medications
  Interventions: Drug: l-arginine

INTERVENTIONS:
Drug: Glutamine — enteral or via NG tube dose of 312mg/kg/day divided every 12 hours from starting feeding + usual care and medications up to 30 says post natal age
  Other Names: Pure a.a. chemical
  Arms: glutamine, PT, sepsis
Drug: l-arginine — enteral or via NG tube dose of 260mg/kg/day divided every 12 hours from starting feeding + usual care and medications up to 30 says post natal age
  Other Names: pure a.a. chemical
  Arms: L-arginine,NEC, PT

SUMMARY:
effects of enteral l-arginine to decrease feeding intolerance and risk of NEC in neonates via its role as a NO precursor. Also, enteral glutamine which may play a role as an immunomodulator on preterm neonates. all these had never been studied in developing countries where sepsis and nec act as a major participant in mortality rates.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is the most common acquired gastrointestinal disease that occurs predominantly in premature infants and is considered to be one of the leading causes of morbidity and mortality in their age group (Schnabl et al., 2008).

Primary prevention of NEC should be the priority, since NEC frequently progresses from nonspecific signs, to extensive necrosis within a matter of hours with medical or surgical treatment, making successful treatment and secondary prevention difficult to achieve (Lin et al., 2013).

One of the assumed novel preventive measures against NEC is L-arginine & glutamine supplementation to high risk infants (Neu, 2005).

We conducted a prospective, interventional, single blinded clinical study in the period from 1/2011- 3/2014 in both NICUs of Children Hospital & Maternity Hospital of Ain Shams University. The study was approved by the Ethical Committee of Faculty of Medicinie, Ain Shams University.

Aim of the study was to assess the preventive role of enteral L-arginine & glutamine against NEC and to assess the role of glutamine in decreasing the impact of sepsis on premature neonates.

Seventy five preterm neonates were enrolled. Inclusion criteria were GA≤ 34 weeks assigned to feed in the first week of life. Exclusion criteria were the presence of any contraindication to feeding (e.g. intestinal surgery), sever or multiple congenital anomalies, intracranial hemorrhage > grade 2 or non- bacterial congenital infection. They were equally divided into 3 groups (L-arginine group, Glutamine group & Control group), 25 neonates per group were randomly enrolled.

L-arginine group included 25 preterm neonates among which 56% were females. Mean for birth weight was 1.45kg, mean for gestational age was 31.84 weeks, 72% were delivered via CS. Median for APGAR score at 1 & 5 minutes were 6 & 8 respectively.

As for the glutamine group, among the 25 neonates included, 52% were females, 92% were born to CS. Mean for birth weight was 1.45kg while mean for GA was 31.84 weeks. Median for APGAR score was 5 in 1st minute (significantly lower than other 2 groups) and 8 at 5 minutes.

In control group that also included 25 neonates, 56% were females and 88% were born to CS. Mean for birth weight was significantly lower if compared to other groups (1.31 kg) while GA was comparable to them (30.64). Median for APGAR score in 1 & 5 minutes was 7 & 8 respectively.

All study subjects received their usual care and medications according to the treating physicians' protocols of management. Additionally, L-arginine group received enteral l-arginine supplementation (starting 0.75mmol/kg/day and reaching 1.5 mmol/kg/day when enteral feeding reaches 40% of full intake), while glutamine group additionally received enteral glutamine supplementations (starting 156mg/kg/day and reaching 312 mg/kg/day when enteral feeding reaches 40% of full intake). The additional enteral supplementations where added with the start of feeding.

Study subjects were followed up daily since the time of enrollment till they were discharged, died or completed 30 days of life. Daily measurement of weight, blood pressure and blood sugar level were done. Feeding protocol of all patients was recorded regarding age on which feeding was initiated, daily increment of feeding, frequency of feeding intolerance, and stoppage of feeding for any stage of NEC. Frequency of septic episodes and hospital stay were also recorded. Plasma l-arginine & glutamine levels were measured at time of enrollment (sample 1), after 15 days of enrollment (sample 2) and at time of diagnosis of any stage of NEC (sample 3). Staging and diagnosis were done according to Bell's criteria. Transcranial ultrasound was done to all study subjects at time of enrollment, before discharge and whenever needed.

Overall incidence of NEC was 12%. Comparing the groups, glutamine group had significant lower incidence of NEC while no difference in NEC incidence was found between L-arginine & control group. Lower gestational age and birth weight were significant risk factors, however; both didn't affect the age of NEC diagnosis. MOD, gender, age on starting feeding and daily increment (wither > 20cc or ≤ 20 cc/kg/day) also didn't affect the incidence of NEC.

Regarding the NEC outcome,3 patients were diagnosed as having NEC in arginine group among which one suffered stage 1 (improved), one suffered stage 2 NEC (improved), and one suffered stage 2 (died), while in control group, among the 6 diagnosed neonates, one suffered stage 1 (died), 5 suffered stage 2 (0ne improved & 4 died). Occurrence of NEC significantly increased risk of mortality & delayed reaching full oral intake.

Overall mortality in the whole study was 13.3%. No significant difference between the 3 groups.

While age on starting feeding was significantly higher in glutamine group (p<0.05), it had no effect on the length of stay or the clinical outcome on the 3 groups. Regarding the frequency of septic episodes, length of stay and attacks of feeding intolerance, no significant difference was reported between the 3 groups.

As for plasma levels of l-arginine & glutamine, no significant difference was estimated among control and glutamine groups regarding initial glutamine levels while edscap group had significantly higher initial l-arginine level compared to l- arginine group. Both l-arginine and glutamine levels were significantly higher in sample 2 in all groups when compared to sample 1 of same patient. However, their levels in sample 2 were significantly correlated to the initial levels rather than their diverse enteral supplementation. No correlation was found between l-arginine and glutamine plasma levels at point of diagnosis of NEC to initial level, gestational age or birth weight. Reaching the full oral intake was significantly delayed in NEC patients, while it wasn't affected by age of initiation of feeding.

Assessing the side effects that may be contributed to L-arginine, incidence of hypotension requiring inotropic management or hyperglycemia requiring insulin therapy showed no statistical significance between the 3 groups denoting possible safety.

Finally, the study supports the finding that enteral glutamine supplementation may be helpful in decreasing the incidence of NEC in preterm neonates. However, this beneficial role was not proven for arginine against NEC, or for glutamine itself against sepsis. Larger studies are needed to confirm the results.

ELIGIBILITY:
Inclusion Criteria:

-Gestational age ≤34 weeks

Exclusion Criteria:

* Severe congenital anomalies.
* Congenital non-bacterial infection
* Evidence of intraventricular hemorrhage (IVH) grade ≥II on cranial ultrasound scan by day 3 of life
* Conjugated hyperbilirubinemia
* Evidence of an inborn error of metabolism
* Exchange transfusion during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-05; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
NEC incidence, stage and outcome | age of 28 days of life
  determining the incidence, stage and outcome of NEC in both l-arginine receiving and control groups

SECONDARY OUTCOMES:
Sepsis | age of 28 days of life
  incidence, severity and outcome of sepsis age at reaching full enteral intake

CONTACTS AND LOCATIONS:
Overall Officials: GHada A. Saleh, MRCPCH, Principal Investigator — Ain Shams University
Locations (1):
- NICU of Children hospital and Nicu of obstetric and gynecology hospital, ain shams university, Cairo, Egypt

REFERENCES:
- [Result] Shah P, Shah V. Arginine supplementation for prevention of necrotising enterocolitis in preterm infants. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD004339. doi: 10.1002/14651858.CD004339.pub3. PMID 17636753
- [Derived] El-Shimi MS, Awad HA, Abdelwahed MA, Mohamed MH, Khafagy SM, Saleh G. Enteral L-Arginine and Glutamine Supplementation for Prevention of NEC in Preterm Neonates. Int J Pediatr. 2015;2015:856091. doi: 10.1155/2015/856091. Epub 2015 Mar 12. PMID 25861285
- See also: Glutamine-enriched enteral nutrition in very low birth weight — http://www.ncbi.nlm.nih.gov/pubmed/15941893
- See also: Arginine supplementation for prevention of necrotising enterocolitis in preterm infants. — http://www.ncbi.nlm.nih.gov/pubmed/15495101